CLINICAL TRIAL: NCT01626625
Title: Mesenchymal Stem Cells; Donor and Role in Management and Reconstruction of Nonunion Fracture
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Ismail Hadisoebroto Dilogo, PhD, Indonesia University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NONUNISTEM1
Record Dates: First submitted 2012-06-12; First posted 2012-06-25 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Healing of Fracture
Keywords: nonunion; stem cells; autograft; hydroxyapatite

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- stem cells (Experimental): stem cells + hydroxy apatite
  Interventions: Drug: stem cells + hydroxy apatite
- autograft (Active Comparator)
  Interventions: Other: autograft taken from iliac crest

INTERVENTIONS:
Drug: stem cells + hydroxy apatite — patient will be transplanted with stem cells and hydroxyapatite
  Arms: stem cells
Other: autograft taken from iliac crest — patient will be transplanted with autograft
  Arms: autograft

SUMMARY:
The investigators hypothesized that mesenchymal stem cells can be isolated from fracture site, iliac crest, and tibial crest, and can be expanded to be used in the management of nonunion fracture.

ELIGIBILITY:
Inclusion Criteria:

* athropic nonunion fracture of the long bone

Exclusion Criteria:

* immunocompromise,
* active infection,
* pathological fracture,
* ongoing hormonal therapy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-04; Primary Completion 2015-04 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
healing of fracture | 1 year
  radiological union

SECONDARY OUTCOMES:
VAS | 1 year
  visual analogue scale

CONTACTS AND LOCATIONS:
Locations (1):
- RSCM, Jakarta, Indonesia